CLINICAL TRIAL: NCT05385510
Title: A Phase Ib Trial to Evaluate the Safety and Immunogenicity of R21/Matrix-M™ in African Children Living With HIV
Brief Title: Assessment of Safety and Immunogenicity of R21/Matrix-M™ in African Children Living With HIV
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: University of Oxford (Other)
Collaborators: MRC/UVRI and LSHTM Uganda Research Unit (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: VAC092
Record Dates: First submitted 2022-05-03; First posted 2022-05-23 (Actual); Last update posted 2024-10-22 (Actual); Status verified 2024-10

CONDITIONS: Malaria
MeSH Terms: conditions — Malaria

STUDY DESIGN:
Intervention Model Description: This is a Phase Ib, open-label, non-randomised, controlled trial. 100 children with confirmed HIV infection will be recruited to group 1. 20 children without HIV infection will be recruited to group 2. All children will receive R21/Matrix-M™
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 - children with HIV (Experimental): 100 5-36 month old children with confirmed HIV infection.
  Interventions: Biological: R21/Matrix-M™
- Group 2 - children without HIV (Experimental): 20 5-36 month old children without HIV infection.
  Interventions: Biological: R21/Matrix-M™

INTERVENTIONS:
Biological: R21/Matrix-M™ — Adjuvanted malaria vaccine

SUMMARY:
A Phase Ib trial to evaluate the safety and immunogenicity of R21/Matrix-M™ in African children living with HIV

DETAILED DESCRIPTION:
This is a Phase Ib, open-label, non-randomised, controlled trial to evaluate the safety and immunogenicity of R21/Matrix-M™ in 5-36 month old African children living with HIV.

The study will be conducted in Uganda at the MRC/UVRI and LSHTM Uganda research unit with recruitment taking place in Kampala, Wakiso and Entebbe.

Children aged 5-36 months will be recruited to the trial. 100 children with confirmed HIV infection will be recruited to group 1. 20 children without HIV infection will be recruited to group 2. Up to 10% variation for each group will be permitted to accommodate variation in the rate of recruitment and retention.

HIV positive children will be recruited from Paediatric HIV care centres within Kampala and Wakiso districts. HIV negative children will be recruited from Entebbe hospital and primary health care centres that provide immunisation and growth monitoring services.

All participants will receive 3 vaccinations of 5µg R21/50µg Matrix-M™. Participants will receive their first dose at 0 months, second dose at 1 month and third dose at 2 months. Participants will receive a booster at 14 months (12 months after their third dose). Participants will be followed up for 12 months following the primary vaccination series and 12 months following the booster dose.

Primary objective:

To assess the safety and reactogenicity profile of the malaria vaccine candidate R21/Matrix-M™ in 5-36-month old African children living with HIV

Secondary objectives:

1. To assess the humoral immunogenicity of R21/Matrix-M™ in 5-36-month-old African children, comparing children living with HIV with HIV negative children
2. To assess the impact of vaccination on HIV reservoir
3. To assess whether increasing age and nadir CD4 count are associated with immunogenicity of R21/Matrix-M™ in 5-36-month-old African children living with HIV

Tertiary objective:

To assess the immunogenicity profile of R21/Matrix-M™ in 5-36-month-old African children, comparing children living with HIV with HIV negative children

This trial is funded by the Serum Institute of India Pvt Ltd.

ELIGIBILITY:
Inclusion Criteria:

* The child must be 5-36 months of age at enrolment (i.e. up to the day of their third birthday).
* Group 1: The child must have HIV infection (documented positive DNA PCR) with WHO stage 1 or 2 HIV disease, whether or not they are receiving ART.
* Group 2: The child must not have HIV infection (absence of HIV infection must be confirmed by documented negative DNA PCR at screening).
* Witnessed, signed/thumb-printed informed consent, obtained from the parent(s)/guardian(s) of the child
* Parents/guardians of the child are able and willing to comply with the requirements of the protocol, in the opinion of the investigator
* The child must be a permanent resident of the study area and likely to remain resident for the duration of the trial.

Exclusion Criteria:

* Previous receipt of a malaria vaccine.
* Enrolment in another malaria intervention trial that could interfere with the results of this study.
* History of severe allergic disease or reactions, including anaphylaxis or angioedema
* History of allergic disease or reactions likely to be exacerbated by any component of the study vaccines, or history of allergic reactions to previous vaccinations
* Clinically significant laboratory abnormality as judged by the study clinician including haemoglobin of ≤8.0 g/dL .
* Major congenital defects.
* Receipt of blood transfusion, immunoglobulins and/or any blood products within the three months preceding enrolment
* Malnutrition requiring hospital admission at the time of enrolment.
* HIV disease of stage 3 or 4, as defined by the WHO clinical staging [23]
* Confirmed or suspected immunosuppressive or immunodeficient state (other than due to HIV infection).

  o This may include asplenia, use of immunosuppressant medication within the past 6 months (except for topical steroids or short-term oral steroids (course lasting <14 days).
* Autoimmune conditions (except mild psoriasis, well-controlled autoimmune thyroid disease, vitiligo or stable coeliac disease)
* Any other clinically significant disease or disorder, or social situation, elicited in medical history, physical examination or laboratory tests that, in the opinion of the study clinician, may:

  * Put the participants at risk because of participation in the trial, or
  * Influence the result of the trial, or
  * Affect the participant's ability to participate in the trial
  * These may include: diseases or disorders of the pulmonary, cardiovascular, gastrointestinal, endocrine, neurological, skin, hepatic or renal systems, cancer, bleeding disorders, abnormalities of screening laboratory tests or examinations
* Receipt of an investigational drug or vaccine other than the study vaccine within 30 days preceding the first dose of study vaccine, or planned use during the study period.
* Current participation in another clinical trial if likely to affect data interpretation of this trial

Ages: 5 Months to 36 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 120 (Estimated)
Dates: Start 2023-01-10 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Solicited local signs and symptoms | 7 days following receipt of each dose
  Occurrence of solicited local signs and symptoms
Solicited systemic signs and symptoms | 7 days following receipt of each dose
  Occurrence of solicited systemic signs and symptoms
SAEs | Through study completion - on average for 15 months
  Occurrence of SAEs
Unsolicited AEs | 30 days following receipt of each dose
  Occurrence of unsolicited adverse events
Clinically significant change from baseline for safety laboratory measures | Through study completion - on average for 15 months
  Clinically significant change from baseline for safety laboratory measures

SECONDARY OUTCOMES:
Antibody responses to CSP and HBsAb | 1 and 6 months following third dose, and 1 and 12 months following booster dose
  Antibody responses to CSP (total anti-IgG responses to NANP and C-term region of CSP) and HBsAb
HIV viral load | 7 days post doses 1 and 2, 30 days post dose 3, and 7, 30 and 365 days post booster
  Change in total HIV DNA copies per million CD4+ T cells
CD4+ count, age at enrolment and vaccine immune response | 1 week after doses 1 and booster, 1 and 6 months after dose 3, and 1 and 12 months after the booster dose
  CD4+ count, age at enrolment and vaccine immune response

OTHER OUTCOMES:
Tertiary - Characterisation of the magnitude and functionality of the cellular and humoral response | Through study completion - on average for 15 months
  Characterisation of the magnitude and functionality of the cellular and humoral response

CONTACTS AND LOCATIONS:
Locations (1):
- MRC/UVRI & LSHTM Uganda Research Unit, Entebbe, Uganda

IPD SHARING:
Plan to Share IPD: Undecided